CLINICAL TRIAL: NCT04351451
Title: Hypomagnesemia and Hypocalcemia Association Following Thyroidectomy
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Amal Abdullah Abdulkareem, consultant&assistant professor, King Saud University
Other Study IDs: 42CFR Part11
Record Dates: First submitted 2020-04-12; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Hypomagnesemia; Hypocalcemia; Hypomagnesemia With Secondary Hypocalcemia
Keywords: Hypomagnesemia; Hypocalcemia; Thyroidectomy
MeSH Terms: conditions — Hypocalcemia; Hypomagnesemia 1, Intestinal | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: thyroidectomy — total thyroidectomy

SUMMARY:
Magnesium plays a role in the active transport of calcium (Ca+2) and potassium ions across cell membranes. Most of it is intracellular or in the bone , however less than 1% of magnesium is in the blood serum. Hypoparathyroidism post thyroidectomy leads to acute Hypocalcemia that leads to hypomagnesemia. The relation of Ca+2 and magnesium (Mg+2) metabolism is complex and mainly related to the interaction of these cations with parathyroid post thyroidectomy. (Mg+2) is an essential regulator of Ca+2 flux and intracellular action of Ca+2. Hypomagnesaemia impairs hypocalcaemia induced PTH release, which is corrected rapidly after magnesium replacement. Attempting to correct only hypocalcemia may prolong symptoms. It is important to monitor both Ca+2 & Mg+2 levels following thyroidectomy to facilitate prompt resolution of symptoms.

Aim of the study: is to highlight the prevalence of hypomagnesemia following thyroidectomy and its association with hypocalcemia which mandate early recognition and treatment to prevent prolongation of hypocalcemia and permanent hypoparathyroidism

Methods:

IRB obtained (E20-4615) informed consent taken from all patient. This is prospective open Label observational study in patients underwent thyroidectomy .the study period was from January 2019 to January 2020. Total of 74 patients with normal renal function. Corrected serum Ca+2, magnesium, phosphate level and vitamin D level are all checked pre operatively and in the first post-operative day.

Result:

Post thyroidectomy 56.8% of patients had hypomagnesemia. 59.5.1% patients had hypocalcemia and 41.9% of patients had low both Ca+2 and Mg+2 (P=0.004)

Conclusion:

Hypocalcemia and hypomagnesemia following thyroidectomy is of multi factorial related mainly to Ca+2, Mg+2 interaction.

Keywords: Hypomagnesemia. Hypocalcemia. Thyroidectomy

DETAILED DESCRIPTION:
Methods:

A prospective study for 1 year starting 1/1/2019 to 1/1/2020. A total 74 patients with normal renal function .admitted for thyroidectomy. Preoperative serum calcium, magnesium, phosphate and vitamin D level all checked. Postoperatively corrected serum calcium, magnesium and phosphate level are checked. The serum calcium less than 2.12mmol/l is corrected with oral or IV calcium infusion plus vitamin D depending on the severity of symptoms. Any serum magnesium less than 0.75mmol/l is corrected with infusion magnesium sulfate. Calcium and magnesium level monitored and corrected according to the result.

Statistical analysis:

Statistical analysis was performed using statistical package for the social sciences (SPSS) version 23.0 software (SPSS Inc., Chicago ,IL,USA). If normal distributed, continuous variable were presented as mean (SD) Student t-test for paired observation was used for statistical. Pearson Chi-square test was used to compare the percentage for categorical variables. P less than 0.05 indicate statistically significant difference

ELIGIBILITY:
Inclusion Criteria:

all patients admitted for thyroidectomy -

Exclusion Criteria:

patient with renal disease

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A prospective study for 1 year starting 1/1/2019 to 1/1/2020. A total 74 patients with normal renal function .admitted for thyroidectomy. Preoperative serum calcium, magnesium, phosphate and vitamin D level all checked. Postoperatively corrected serum calcium, magnesium and phosphate level are checked. The serum calcium less than 2.12mmol/l is corrected with oral or IV calcium infusion plus vitamin D depending on the severity of symptoms. Any serum magnesium less than 0.75mmol/l is corrected with infusion magnesium sulfate. Calcium and magnesium level monitored and corrected according to the result.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
hypomagnesemia post thyroidectomy | one year period
  magnesium serum level less than 0.75 mmol/l
Hypocalcemia post thyroidectomy | one year period
  calcium serum level less than 2.12 mmol/l

SECONDARY OUTCOMES:
association of Hypomagnesemia and Hypocalcemia | one year period
  calculate the percentage of association of both metabolic derangement post thyroidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine , King Saud University, Riyadh, Central Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No